CLINICAL TRIAL: NCT04552873
Title: Urea Therapy for Hyponatremia in Subarachnoid Hemorrhage
Acronym: NAT-URE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 38RC19.189
Record Dates: First submitted 2020-09-10; First posted 2020-09-17 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Hyponatremia; Subarachnoid Hemorrhage; SIADH
Keywords: urea; copeptine; hyponatremia; SAH; SIADH
MeSH Terms: conditions — Hyponatremia; Subarachnoid Hemorrhage; Inappropriate ADH Syndrome | interventions — Urea

STUDY DESIGN:
Intervention Model Description: Comparative study in 2 parallel arms, monocentric, randomized, double blind.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): the experimental group will be treated during 5 days by urea dose per administration : 1g / kg / 24 hours in 2 or 3 doses morning, noon and evening (dose adjustment of urea according to weight)
  Interventions: Drug: Urea
- CONTROL GROUP (Placebo Comparator): the control group will be treated during 5 days by ergytonyl dose per administration : 5mL
  Interventions: Other: PLACEBO

INTERVENTIONS:
Drug: Urea — the experimental group will be treated during 5 days by urea dose per administration : 1g / kg / 24 hours in 2 or 3 doses morning, noon and evening (dose adjustment of urea according to weight)
  If hyponatremia persists beyond D8 after initiation of the study treatment (urea or placebo), that is to say after the date of the collection of the primary endpoint, it will be possible to introduce corticosteroids (fludrocortisone or others). These treatments will be collated.
  If during patient monitoring the serum sodium exceeds 145 mmol / L, treatment should no longer be administered.
  Arms: EXPERIMENTAL GROUP
Other: PLACEBO — the control group will be treated during 5 days by ergytonyl dose per administration : 5mL
  Arms: CONTROL GROUP

SUMMARY:
Hyponatremia is defined as a plasma sodium concentration below 135 mmol / L. This is a common occurrence (20-50%) during subarachnoid hemorrhage (SAH). Its appearance is often associated with vasospasm. It is associated with an increase in morbidity and mortality linked to induced neurological disorders. Hyponatremia is caused by two etiologies: the syndrome of inappropriate secretion of anti-diuretic hormone (SIADH), and the cerebral salt wasting syndrome, CSWS. Theoretically, these two entities are differentiated by the patient's volemia; in practice, this parameter is difficult to measure. In addition, the correction of hyponatremia is diametrically opposed according to its mechanism: water restriction in the case of SIADH, sodium intake in the event of CSWS. Urea is offered as a second-line treatment in the event of treatment failure to correct hyponatremia. However, the efficacy of this treatment is based on small, observational, retrospective studies. Moreover, the mechanism of action of urea remains poorly understood: it could be a hyperosmolar effect or passive renal reabsorption of sodium.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged at least 18 years old
* Non-traumatic HSA
* Hyponatremia defined by a natremia less than 135 mmol / L and a high natriuresis, greater than 250 mmol / L despite well-managed saline intakes

Exclusion Criteria:

* Severe cardiac decompensation (LVEF <30%)
* Severe hepatic cirrhosis (PT <30%, ascites), known severe renal failure (GFR <30mL / min / 1.73m²)
* Blood urea> 25 mmol / L in the basal state
* Osmotherapy and diuretics in the last 48 hours
* Ongoing treatment with systemic corticosteroids
* Persons referred to in Articles L1121-5 to L1121-8 of the CSP corresponding to all protected persons: pregnant woman, parturient, nursing mother, person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure.
* Patient not affiliated to a social security scheme
* Known hypersensitivity to any of the components of ergytonyl
* Contraindications to ergytonyl: taking curative anticoagulants, previously known and treated diabetic patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the effectiveness of urea therapy in correcting persistent hyponatremia despite adequate management during subarachnoid hemorrhage | 5 days
  Change in blood serum in mmol / L measured before initiation of treatment and on the day of discontinuation of treatment

SECONDARY OUTCOMES:
To compare the sodium intake required to correct the natremia. | 8 days
  Measurement of daily sodium intake in each group
To study the mechanism of action of urea | 48 hours after the end of treatment
  Daily plasma co-peptin levels in each group during treatment and 48 hours after cessation of treatment.
To assess the impact of treatment on length of stay | 3 months
  Length of stay in intensive care and/or continuing care unit
To assess the impact of treatment on neurological outcome at 3 months from inclusion | 3 months
  Measurement of modified Rankin score
To assess the adverse effects of treatment | 3 months
  Prevalence of adverse effects of urea (headaches, digestive disorders, etc.)
Persistence of correction of natraemia 48H after cessation of treatment | 48 hours after the end of treatment
  Variation in natraemia mmol/L measured before introduction of treatment and 48 hours after cessation of treatment
To compare the speed of correction of natraemia | 5 days
  Average time taken for natraemia to correct to Na > 135 mmol/L after initiation of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Perrine BOUCHEIX, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hall A, O'Kane R. The Extracranial Consequences of Subarachnoid Hemorrhage. World Neurosurg. 2018 Jan;109:381-392. doi: 10.1016/j.wneu.2017.10.016. Epub 2017 Oct 16. PMID 29051110
- [Background] Mapa B, Taylor BE, Appelboom G, Bruce EM, Claassen J, Connolly ES Jr. Impact of Hyponatremia on Morbidity, Mortality, and Complications After Aneurysmal Subarachnoid Hemorrhage: A Systematic Review. World Neurosurg. 2016 Jan;85:305-14. doi: 10.1016/j.wneu.2015.08.054. Epub 2015 Sep 7. PMID 26361321
- [Background] Hannon MJ, Behan LA, O'Brien MM, Tormey W, Ball SG, Javadpour M, Sherlock M, Thompson CJ. Hyponatremia following mild/moderate subarachnoid hemorrhage is due to SIAD and glucocorticoid deficiency and not cerebral salt wasting. J Clin Endocrinol Metab. 2014 Jan;99(1):291-8. doi: 10.1210/jc.2013-3032. Epub 2013 Dec 20. PMID 24248182
- [Background] Nakajima H, Okada H, Hirose K, Murakami T, Shiotsu Y, Kadono M, Inoue M, Hasegawa G. Cerebral Salt-wasting Syndrome and Inappropriate Antidiuretic Hormone Syndrome after Subarachnoid Hemorrhaging. Intern Med. 2017;56(6):677-680. doi: 10.2169/internalmedicine.56.6843. Epub 2017 Mar 17. PMID 28321069
- [Background] Hoorn EJ, Zietse R. Diagnosis and Treatment of Hyponatremia: Compilation of the Guidelines. J Am Soc Nephrol. 2017 May;28(5):1340-1349. doi: 10.1681/ASN.2016101139. Epub 2017 Feb 7. PMID 28174217